CLINICAL TRIAL: NCT05781542
Title: A Phase-1 Open-label Clinical Trial to Evaluate the Safety and Immunogenicity of Synthetic DNAs Encoding NP-GT8 and IL-12, With or Without a TLR-agonist- Adjuvanted HIV Env Trimer 4571 Boost, in Adults Without HIV
Brief Title: Clinical Trial to Evaluate the Safety and Immunogenicity of Synthetic DNAs Encoding NP-GT8 and IL-12, With or Without a TLR-agonist-Adjuvanted HIV Env Trimer 4571 Boost, in Adults Without HIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: HIV Vaccine Trials Network (Network); The Wistar Institute (Other); The Betty and Dale Bumpers Vaccine Research Center (VRC) (Unknown); Inovio Pharmaceuticals (Industry); Access to Advanced Health Institute (AAHI) (Other); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 305
Record Dates: First submitted 2023-01-11; First posted 2023-03-23 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — aluminum sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): a total of approximately 9 participants will receive 3 administrations of sD-NP-GT8 DNA at a dose of 0.4 mg, coformulated with IL-12 DNA at a dose of 0.1 mg at days 1, 29, and 85. Study products will be administered intradermally via EP of the skin on each upper arm
  Interventions: Biological: sD-NP-GT8 DNA; Biological: IL-12 DNA
- Group 2 (Experimental): a total of approximately 18 participants will receive 3 administrations of sD-NP-GT8 DNA at a dose of 1.6 mg, coformulated with IL-12 DNA at a dose of 0.4 mg at days 1, 29, and 85. Study products will be administered intradermally via EP of the skin on each upper arm
  Interventions: Biological: sD-NP-GT8 DNA; Biological: IL-12 DNA
- Group 3 (Experimental): a total of approximately 18 participants will receive 3 administrations of sD-NP-GT8 DNA at a dose of 1.6 mg, coformulated with IL-12 DNA at a dose of 0.4 mg at days 1, 29, and 85. These doses will be administered intradermally via EP of the skin on each upper arm. All participants in Group 3 will also receive 2 administrations of Trimer 4571 at a dose of 100 mcg adjuvanted with 5 mcg of 3M-052-AF + 500 mcg Alum via IM injections into the deltoid muscle at days 85 and 169
  Interventions: Biological: sD-NP-GT8 DNA; Biological: IL-12 DNA; Biological: Trimer 4571; Biological: 3M-052-AF; Drug: Alum

INTERVENTIONS:
Biological: sD-NP-GT8 DNA — 0.4 mg
  Arms: Group 1
Biological: sD-NP-GT8 DNA — 1.6 mg
  Arms: Group 2; Group 3
Biological: IL-12 DNA — 0.1 mg
  Arms: Group 1
Biological: IL-12 DNA — 0.4 mg
  Arms: Group 2; Group 3
Biological: Trimer 4571 — 100 mcg
  Arms: Group 3
Biological: 3M-052-AF — 5 mcg
  Arms: Group 3
Drug: Alum — 500 mcg
  Arms: Group 3

SUMMARY:
This is an open-label study to examine the safety and immunogenicity of synthetic DNAs encoding NP-GT8 and IL-12 with or without a TLR-agonist-adjuvanted Env Trimer 4571 boost in adults without HIV. The primary hypothesis is that vaccination with this recombinant DNA vaccine encoding a germline-targeting epitope followed by a trimeric protein boost will elicit VRC01-class B-cell responses as well as antigen-specific T-cell responses.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to complete the informed consent process, including an Assessment of Understanding (AoU): volunteer demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly.
* 18 to 55 years old, inclusive, on day of enrollment.
* Available for clinic follow-up through the last clinic visit and willing to be contacted at least 12 months after the last vaccine administration.
* Willing to undergo leukapheresis.
* Agrees not to enroll in another study of an investigational agent during participation in the trial.
* In good general health according to the clinical judgement of the site investigator.
* Physical examination and laboratory results without clinically significant findings that would interfere with assessment of safety or reactogenicity in the clinical judgement of the site investigator.
* Assessed as low risk for HIV acquisition per low-risk guidelines, agrees to discuss HIV-infection risks, agrees to risk-reduction counseling, and agrees to avoid behaviors associated with high risk of HIV exposure through the final study visit. Low risk may include persons stably taking HIV pre-exposure prophylaxis (PrEP) as prescribed for 6 months or longer.
* Hemoglobin:

  * ≥ 11.0 g/dL for volunteers who were assigned female sex at birth.
  * ≥ 13.0 g/dL for volunteers who were assigned male sex at birth and transgender males who have been on hormone therapy for more than 6 consecutive months.
  * ≥ 12.0 g/dL for transgender females who have been on hormone therapy for more than 6 consecutive months.
  * For transgender participants who have been on hormone therapy for less than 6 consecutive months, determine hemoglobin eligibility based on the sex assigned at birth.
* Platelets = 125,000-550,000/mm3
* White blood cell (WBC) count = 2,500-12,000/mm3 (not exclusionary: if count greater than 12,000 with investigation showing general good health and PSRT approval). The Leukapheresis Center may impose a higher lower limit of 3,500/mm3
* Alanine aminotransferase (ALT) < 2.5 x upper limit of normal (ULN) based on the institutional normal range.
* Serum creatinine ≤ 1.1 x ULN based on the institutional normal range.
* Corrected total serum calcium level of > 8.5 mg/dL.
* Blood pressure in the range of 90 to < 140 mmHg systolic and 50 to < 90 mmHg diastolic.
* Negative results for HIV infection by a US Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA) or chemiluminescent microparticle immunoassay (CMIA).
* Negative for anti-Hepatitis C Abs (anti-HCV), or negative HCV nucleic acid test (NAT) if anti-HCV Abs are detected.
* Negative for Hepatitis B surface antigen.
* For a volunteer capable of becoming pregnant:

  * Volunteers who were assigned female sex at birth and are of reproductive potential must agree to use effective means of birth control from at least 21 days prior to enrollment through 8 weeks after their last vaccination timepoint.
  * Has negative beta human chorionic gonadotropin (β-HCG) pregnancy test (urine or serum) on day of enrollment.

Exclusion Criteria:

* Volunteer who is breast-feeding or pregnant.
* Morbid obesity. Enrollment of individuals with body mass index (BMI) that is

  ≥ 40, whom the site investigator assesses are in good health, may be considered by PSRT on a case-by-case basis.
* Diabetes mellitus (DM). Type 2 DM, controlled with diet alone, or a history of isolated gestational diabetes are not exclusionary. Enrollment of individuals with Type 2 DM that is well-controlled on hypoglycemic agent(s) may be considered, provided the HgbA1c is ≤ 8% within the last 6 months (sites may draw these at screening).
* Previous or current recipient of an investigational HIV vaccine (previous placebo recipients are not excluded).
* Systemic glucocorticoid use equal to or greater than prednisone 10 mg/day within 3 months prior to enrollment, congenital or acquired immunodeficiency, or other systemic medication use likely to impair immune response to vaccine in the opinion of the site investigator.
* Blood products or immunoglobulin within 16 weeks prior to enrollment; receipt of immunoglobulin within 16 weeks prior to enrollment requires PSRT approval.
* Receipt of any live attenuated vaccine within 4 weeks prior to enrollment. (Note: ACAM2000 vaccine for Monkeypox received within 30 days prior to enrollment or receipt of study vaccine, or if ACAM2000 received greater than 30 days prior to enrollment, or prior to receipt of study vaccine and vaccination scab still present; or planned administration within 30 days after enrollment or receipt of study vaccine).
* Receipt of any vaccines that are not live attenuated within 14 days prior to enrollment; replication incompetent vaccines such as the Jynneos vaccine for the prevention of monkeypox disease are not considered to be live vaccines.
* Non-HIV experimental vaccine(s) received within the last 1 year in a prior vaccine trial. Exceptions may be made by the HVTN 305 PSRT for vaccines that have subsequently undergone licensure or Emergency Use Authorization by the FDA or, if outside the United States, equivalent authorization by the national regulatory authority.
* Initiation of antigen-based immunotherapy for allergies within the previous year (stable immunotherapy is not exclusionary); inclusion of participants who initiated immunotherapy within the previous year requires PSRT approval.
* Receipt of investigational research agents with a half-life of 7 or fewer days within 4 weeks prior to enrollment. If a potential participant has received investigational agents with a half-life greater than 7 days (or unknown half-life) within the past year, PSRT approval is required for enrollment.
* Serious reactions to vaccines that preclude receipt of study injections as determined by the principal investigator (PI) or designee, including history of serious reaction (eg, hypersensitivity, anaphylaxis) to any or any component of the study vaccine.
* Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema.
* Idiopathic urticaria within the past year.
* Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions).
* Seizure disorder; febrile seizures as a child or seizures secondary to alcohol withdrawal more than 5 years ago are not exclusionary.
* Asplenia or functional asplenia.
* Active duty and reserve US military personnel.
* Any other chronic or clinically significant condition that in the clinical judgement of the investigator would jeopardize the safety or rights of the study participant, including, but not limited to: clinically significant forms of drug or alcohol abuse, serious psychiatric disorders, persons with any suicide attempt within the past one year (if between 1-2 years, consult PSRT) or cancer that, in the clinical judgment of the site investigator, has a potential for recurrence (excluding basal cell carcinoma).
* Asthma is excluded if the participant has ANY of the following:

  * Required either oral or parenteral corticosteroids for an exacerbation two or more times within the past year; OR
  * Required either oral or parenteral corticosteroids for an exacerbation 2 or more times within the past year; OR
  * Needed emergency care, urgent care, hospitalization, or intubation for an acute asthma exacerbation within the past year (eg, would NOT exclude individuals with asthma who meet all other criteria but sought urgent/emergent care solely for asthma medication refills or coexisting conditions unrelated to asthma); OR
  * Uses a short-acting rescue inhaler more than 2 days per week for acute asthma symptoms (ie, not for preventive treatment prior to athletic activity); OR
  * Uses medium-to-high-dose inhaled corticosteroids (greater than 250 mcg fluticasone or therapeutic equivalent per day), whether in single-therapy or dual-therapy inhalers (ie, with a long-acting beta agonist [LABA]); OR
  * Uses more than 1 medication for maintenance therapy daily. Inclusion of anyone on a stable dose of more than 1 medication for maintenance therapy daily for greater than 2 years requires PSRT approval.
* A participant with a history of an immune-mediated disease, either active or remote. Specific examples are listed in Appendix I (AESI index). Not exclusionary: 1) remote history of Bell's palsy (>2 years ago) not associated with other neurologic symptoms, 2) mild psoriasis that does not require ongoing systemic treatment.
* History of allergy to local anesthetic (Novocaine, Lidocaine).
* Investigator concern for difficulty with venous access based upon clinical history and physical examination. For example, history of IV drug abuse or substantial difficulty with previous blood draws.
* Presence of implanted electronic medical device (eg, pacemaker, implantable cardioverter defibrillator).
* Presence of surgical or traumatic metal implant in either upper arm and/or upper torso.
* History of cardiac arrhythmia (eg, supraventricular tachycardia, atrial fibrillation) (Not excluded: sinus arrhythmia).
* Tattoo overlying the injection sites preventing assessment of reactogenicity in the view of the investigator or skin condition at the injection sites.
* History or presence of keloid scar formation or hypertrophic scar

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2025-04-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (4):
  - Alabama CRS (Site ID: 31788), Birmingham, Alabama
  - Bridge HIV CRS, San Francisco, California
  - San Francisco Vaccine and Prevention CRS, San Francisco, California
  - Brigham and Women's Hospital Vaccine CRS [30007], Boston, Massachusetts
- South Africa (4):
  - Soweto HVTN CRS, Johannesburg, Gauteng
  - CAPRISA eThekwini CRS, Durban, KwaZulu-Natal
  - Durban Adult HIV CRS, Durban, KwaZulu-Natal
  - Groote Schuur HIV CRS (Site ID: 31708), Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group T1: 0.5mg INO-6172 (m0,1,3)
- Group T2: 2mg INO-6172 (m0,1,3)
- Group T3: 2mg INO-6172 (m0,1,3), 100mcg Trimer 4571 + 5mcg 3M-052 AF/500 mcg Alum (m3,6)
Period: Overall Study
Arm/Group | Group T1 | Group T2 | Group T3
Started | 10 | 18 | 18
Safety Population | 10 | 18 | 18
Completed | 9 | 18 | 17
Not Completed | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group T1 | Group T2 | Group T3 | Total
Number analyzed (Participants) | 10 | 18 | 18 | 46
Age, Continuous [Median (Full Range); unit: years] | 28 [20 to 53] | 25.5 [20 to 43] | 24 [18 to 51] | 25 [18 to 53]
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years | 0 | 0 | 0 | 0
  18 - 20 years | 1 | 1 | 4 | 6
  21 - 30 years | 5 | 12 | 10 | 27
  31 - 40 years | 3 | 4 | 3 | 10
  41 - 50 years | 0 | 1 | 0 | 1
  Above 50 years | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 6 | 18
  Male | 6 | 10 | 12 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 5
  Not Hispanic or Latino | 9 | 16 | 16 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 14 | 10 | 27
  White | 7 | 4 | 6 | 17
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 3 | 14 | 9 | 26
  United States | 7 | 4 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Solicited Adverse Events Signs and Symptoms: Pain and/or Tenderness
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The maximum grade observed for each symptom over the time frame is presented
Time Frame: Measured through 7 days following vaccine administration for INO-6172 alone and 14 days following vaccine administration for Trimer 4571 + 3M-052-AF/Alum
Population: Started (enrolled).
Measure: Count of Participants; unit: Participants
Arm/Group | Group T1 | Group T2 | Group T3
Number analyzed (Participants) | 10 | 18 | 18
Participants
  None | 3 | 9 | 4
  Mild | 6 | 8 | 10
  Moderate | 1 | 1 | 1
  Severe | 0 | 0 | 3
  Potentially Life-threatening | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Local Solicited Adverse Events Signs and Symptoms: Erythema and/or Induration
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Started (enrolled).
Measure: Count of Participants; unit: Participants
Arm/Group | Group T1 | Group T2 | Group T3
Number analyzed (Participants) | 10 | 18 | 18
Participants
  Erythema/Redness: None | 8 | 13 | 13
  Erythema/Redness: Mild | 1 | 4 | 5
  Erythema/Redness: Moderate | 1 | 1 | 0
  Erythema/Redness: Severe | 0 | 0 | 0
  Erythema/Redness: Potentially Life-threatening | 0 | 0 | 0
  Induration/Swelling: None | 8 | 16 | 16
  Induration/Swelling: Mild | 2 | 2 | 2
  Induration/Swelling: Moderate | 0 | 0 | 0
  Induration/Swelling: Severe | 0 | 0 | 0
  Induration/Swelling: Potentially Life-threatening | 0 | 0 | 0
  Erythema and/or Induration: None | 8 | 13 | 13
  Erythema and/or Induration: Mild | 1 | 4 | 5
  Erythema and/or Induration: Moderate | 1 | 1 | 0
  Erythema and/or Induration: Severe | 0 | 0 | 0
  Erythema and/or Induration: Potentially Life-threatening | 0 | 0 | 0

3. Primary Outcome: Number of Participants Reporting Unsolicited Adverse Events (AEs), by Severity Grade
Description: The number (percentage) of Participants Reporting Unsolicited Adverse Events (AEs) was summarized by arm and severity grade. The number (percentage) of Participants Reporting Unsolicited Adverse Events (AEs) was summarized by arm and severity grade. Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 (exceptions apply)
Time Frame: as for outcome 1
Population: Started (enrolled).
Measure: Count of Participants; unit: Participants
Arm/Group | Group T1 | Group T2 | Group T3
Number analyzed (Participants) | 10 | 18 | 18
Participants
  Malaise and/or fatigue: None | 7 | 10 | 4
  Malaise and/or fatigue: Mild | 2 | 5 | 5
  Malaise and/or fatigue: Moderate | 1 | 2 | 4
  Malaise and/or fatigue: Severe | 0 | 1 | 5
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0 | 0
  Myalgia: None | 9 | 13 | 5
  Myalgia: Mild | 1 | 5 | 7
  Myalgia: Moderate | 0 | 0 | 2
  Myalgia: Severe | 0 | 0 | 4
  Myalgia: Potentially Life-threatening | 0 | 0 | 0
  Headache: None | 7 | 11 | 5
  Headache: Mild | 2 | 4 | 7
  Headache: Moderate | 1 | 2 | 1
  Headache: Severe | 0 | 1 | 5
  Headache: Potentially Life-threatening | 0 | 0 | 0
  Nausea: None | 9 | 14 | 9
  Nausea: Mild | 1 | 3 | 6
  Nausea: Moderate | 0 | 1 | 3
  Nausea: Severe | 0 | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0 | 0
  Chills: None | 10 | 14 | 5
  Chills: Mild | 0 | 4 | 8
  Chills: Moderate | 0 | 0 | 2
  Chills: Severe | 0 | 0 | 3
  Chills: Potentially Life-threatening | 0 | 0 | 0
  Arthralgia: None | 9 | 16 | 7
  Arthralgia: Mild | 1 | 2 | 5
  Arthralgia: Moderate | 0 | 0 | 4
  Arthralgia: Severe | 0 | 0 | 2
  Arthralgia: Potentially Life-threatening | 0 | 0 | 0
  Max. Systemic Symptoms: None | 6 | 9 | 3
  Max. Systemic Symptoms: Mild | 3 | 4 | 5
  Max. Systemic Symptoms: Moderate | 1 | 4 | 3
  Max. Systemic Symptoms: Severe | 0 | 1 | 7
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0 | 0
  Temperature: None | 10 | 17 | 13
  Temperature: Mild | 0 | 1 | 3
  Temperature: Moderate | 0 | 0 | 2
  Temperature: Severe | 0 | 0 | 0
  Temperature: Potentially Life-threatening | 0 | 0 | 0

4. Primary Outcome: Number of Participants Reporting Unsolicited Adverse Events (AEs), by Severity Grade
Description: The number (percentage) of Participants Reporting Unsolicited Adverse Events (AEs) was summarized by arm and severity grade. Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 (exceptions apply)
Time Frame: Measured for 30 days after any receipt of study vaccination
Population: Started (enrolled).
Measure: Count of Participants; unit: Participants
Arm/Group | Group T1 | Group T2 | Group T3
Number analyzed (Participants) | 10 | 18 | 18
Participants
  Mild | 0 | 2 | 3
  Moderate | 5 | 6 | 9
  Severe | 0 | 0 | 1
  Potentially life-threatening | 0 | 0 | 0

5. Primary Outcome: Number of Participants Reporting Medically Attended Adverse Events (MAAEs), by Severity Grade
Description: The number (percentage) of Participants Reporting Medically Attended Adverse Events (MAAEs) was summarized by arm and severity grade
Time Frame: Measured through Month 12 following any receipt of study products
Population: Started (enrolled).
Measure: Count of Participants; unit: Participants
Arm/Group | Group T1 | Group T2 | Group T3
Number analyzed (Participants) | 10 | 18 | 18
Participants
  Mild | 0 | 0 | 0
  Moderate | 5 | 4 | 7
  Severe | 0 | 0 | 0
  Potentially life-threatening | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Early Discontinuation of Vaccinations and Reason for Discontinuation
Description: The number (percentage) of participants with early discontinuation of vaccinations and reason for discontinuation was summarized by arm
Time Frame: Measured through Month 12 following any receipt of study products
Population: Started (enrolled).
Measure: Count of Participants; unit: Participants
Arm/Group | Group T1 | Group T2 | Group T3
Number analyzed (Participants) | 10 | 18 | 18
Participants
  Unable to contact participant | 1 | 0 | 0
  Protocol deviation | 0 | 1 | 0
  Did not discontinue SPA | 9 | 17 | 18

7. Primary Outcome: Number of Participants With Early Study Termination and Reason for Early Study Termination
Description: The number (percentage) of participants with early study termination and reason for early study termination was summarized by arm
Time Frame: Measured through Month 12 following any receipt of study products
Population: Started (enrolled).
Measure: Count of Participants; unit: Participants
Arm/Group | Group T1 | Group T2 | Group T3
Number analyzed (Participants) | 10 | 18 | 18
Participants
  Unable to contact participant | 1 | 0 | 1
  Scheduled exit visit/end of study | 9 | 18 | 17

ADVERSE EVENTS:
Time Frame: The AE reporting period for this study comprises the entire study period for each individual participant (from the participant's study enrollment until his or her study completion or discontinuation), up to 18 months.
Description: The number (percentage) of Participants Reporting Solicited AEs and unsolicited AEs including All-Cause Mortality, Serious Adverse Events (SAEs), and Other (Not Including Serious) Adverse Events were summarized by arm
Arm/Group | Group T1 | Group T2 | Group T3
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 8/10 | 14/18 | 17/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group T1 (N=10) | Group T2 (N=18) | Group T3 (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Solicited) (Gastrointestinal disorders) | 1 (1) | 4 (4) | 9 (9)
Chills (Solicited) (General disorders) | 0 (0) | 4 (4) | 13 (13)
Cyst (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (Solicited) (General disorders) | 2 (2) | 5 (5) | 5 (5)
Injection site pain (Solicited) (General disorders) | 7 (7) | 9 (9) | 14 (14)
Injection site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site swelling (Solicited) (General disorders) | 2 (2) | 2 (2) | 2 (2)
Malaise (Solicited) (General disorders) | 3 (3) | 8 (8) | 14 (14)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Norovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal gonococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (4)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Syphilis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Body temperature increased (Solicited) (Investigations) | 0 (0) | 1 (1) | 5 (5)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 2 (3)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Solicited) (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 11 (11)
Myalgia (Solicited) (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 13 (13)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Solicited) (Nervous system disorders) | 3 (3) | 7 (7) | 13 (13)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Victim of sexual abuse (Social circumstances) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/42/NCT05781542/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT05781542/SAP_001.pdf